CLINICAL TRIAL: NCT05966961
Title: 'All Comer'/'Real-world' Registry-based Randomized, Prospective, Multicenter Clinical Trial to Evaluate the Incidence of Complications Using Novosyn® CHD Suture Versus Polyglactin 910 Suture to Close the Wound After Emergency or Elective Laparotomy or Laparoscopic Surgery
Brief Title: Novosyn® CHD vs Polyglactin 910 Suture to Close Wounds After Emergency or Elective Laparotomy or Laparoscopic Surgery
Acronym: POLYNOVO-CHD
Status: Recruiting | Type: Observational
Sponsor: Aesculap AG (Industry)
Collaborators: B.Braun Surgical SA (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-G-H-2201
Record Dates: First submitted 2023-07-19; First posted 2023-08-01 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Surgical Site Infection
Keywords: Chlorhexidine coated suture; emergency laparoscopic surgery; emergency laparotomy surgery; elective laparoscopic surgery; elective laparotomy surgery; Novosyn®; Polyglactin 910
MeSH Terms: conditions — Surgical Wound Infection | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Novosyn®: Sutures will be used to close the laparotomy or trocar incision in emergency or elective surgery. The suture material will be applied for fascia closure (and subcutaneous closure if applicable) in the context of daily clinical routine
  Interventions: Device: Novosyn® in emergency or elective laparotomy or laparoscopic surgery
- Polyglactin 910: Sutures will be used to close the laparotomy or trocar incision in emergency or elective surgery. The suture material will be applied for fascia closure (and subcutaneous closure if applicable) in the context of daily clinical routine
  Interventions: Device: Polyglactin 910 in emergency or elective laparotomy or laparoscopic surgery

INTERVENTIONS:
Device: Novosyn® in emergency or elective laparotomy or laparoscopic surgery — Fascia closure (and subcutaneous closure if applicable) after emergency or elective laparotomy or laparoscopic surgery.
  Groups: Novosyn®
Device: Polyglactin 910 in emergency or elective laparotomy or laparoscopic surgery — Fascia closure (and subcutaneous closure if applicable) after emergency or elective laparotomy or laparoscopic surgery.
  Groups: Polyglactin 910

SUMMARY:
The aim of the study is to elucidate, if the colonization of bacteria is lower on the Novosyn® CHD suture compared to uncoated Polyglactin 910 suture, which will be assessed by the incidence of surgical site infections (SSI: A1 and A2). The results of this registry will generate further clinical evidence for the use and the benefit of a Chlorhexidine coated suture used to close the wound after an emergency or elective laparoscopic or laparotomy surgery. The benefit for individual patients lies in the early diagnosis of complications and in the optimized postoperative controls of a clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing an emergency or elective laparotomy or laparoscopic surgery.
* Written informed consent
* Age≥ 18 years
* Not incapacitated patient

Exclusion Criteria:

* No exclusion criteria except patients with allergy or hypersensitivity to chlorhexidine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing wound closure after emergency or elective laparoscopic or laparotomy surgery
Sampling Method: Probability Sample
Enrollment: 2998 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Frequency of surgical site infection (superficial (A1) and deep (A2) | until 30 days + 5 days after surgery.
  The aim of the study is to elucidate, if the colonization of bacteria is lower on the Novosyn® CHD suture compared to uncoated Polyglactin 910 suture, which will be assessed by the incidence of surgical site infections (SSI: A1 and A2).

SECONDARY OUTCOMES:
Handling of the suture material | intraoperatively
  Assessment of the handling of the suture material intraoperatively using a questionnaire including different dimensions (knot security, tensile strength, knot run down, tissue drag etc.) with 5 evaluations levels (excellent, very good, good, satisfied, poor).
Length of hospital stay | until discharge (approximately 10 days after surgery)
  Number of days the patient has to stay in hospital after emergency or elective laparotomy or laparoscopic surgery
Time to return to work | until 30 days + 5 days after surgery.
  Number of days the patient needed to return to work after emergency or elective laparotomy or laparoscopic surgery
Incidence of Surgical Site Infection (SSI) | at discharge (approximately 10 days after surgery)
  Incidence of Surgical Site Infection (SSI) (superficial (A1), deep (A2) and organ space (A3)) at the time of discharge
Incidence of SSI (superficial (A1), deep (A2) and organ space (A3)) stratified by wound class | until 30 days + 5 days after surgery
  Incidence of SSI (superficial (A1), deep (A2) and organ space (A3)) stratified by wound class (Class I clean, Class II clean/contaminated, Class III contaminated, Class IV dirty/infected)
Cumulative Rate of postoperative complications | discharge (approximately 10 days after surgery) and 30 days+ 5 days after surgery.
  Number of postoperative complications of any kind for descriptive analysis
Cumulative Rate of reoperation | at discharge (approximately 10 days after surgery) and 30 days + 5 days after surgery.
  Number of reoperation of any kind for descriptive analysis
Cumulative Rate of suture removal due to wound problems | at discharge (approximately 10 days after surgery) and 30 days + 5 days after surgery.
  Rate of suture removal due to wound problems (infection, dehiscence, residual material requiring removal) for descriptive analysis
Cumulative Rate of Re-suturing | at discharge (approximately 10 days after surgery) and 30 days + 5 days after surgery.
  Rate of Re-suturing of any kind for descriptive analysis
Hernia rate | 30 days + 5 days postoperatively
  Number of Wound Hernia including umbilical hernia verified by ultra-sound examination

CONTACTS AND LOCATIONS:
Overall Officials: Antonio José Torres Garcia, Prof. Dr., Principal Investigator — Hospital San Carlos, Madrid
Locations (4):
- Pineta Grande Hospital, Napoli, Italy
- Spain (3):
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital Universitario Virgen del Rocío, Seville

IPD SHARING:
Plan to Share IPD: No